CLINICAL TRIAL: NCT01870570
Title: Determination of Glycaemic Index and Insulinaemic Index Values of 6 Cereal Products in 3 Separate Research Centers
Brief Title: Determination of Glycaemic Index and Insulinaemic Index Values of 6 Food Products in 3 Separate Research Centers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mondelēz International, Inc. (Industry)
Collaborators: BioFortis (Other); Glycemic Index Laboratories, Inc (Industry); University of Sydney (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: KBE019
Record Dates: First submitted 2013-06-03; First posted 2013-06-06 (Estimated); Last update posted 2014-08-21 (Estimated); Status verified 2014-08

CONDITIONS: Glycaemia; Insulinemia
Keywords: Glycaemia; Insulinemia
MeSH Terms: interventions — Glucose

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (7):
- Reference Glucose (Other): Glucose Standard (50g of Glucose)
  Interventions: Other: Reference Glucose
- Food Product A: Corn Flakes (Experimental): Corn Flakes
  Interventions: Other: Food Product A: Corn Flakes
- Food Product B: Ginger Bread (Experimental): Ginger Bread
  Interventions: Other: Food Product B: Ginger Bread
- Food Product C:Sandwiched Breakfast Biscuit (Experimental): Sandwiched Breakfast Biscuit
  Interventions: Other: Food Product C:Sandwiched Breakfast Biscuit
- Food Product D: Crackers Nature (Experimental): Crackers Nature
  Interventions: Other: Food Product D: Crackers Nature
- Food Product E: Breakfast Biscuit (Experimental): Breakfast Biscuit
  Interventions: Other: Food Product E: Breakfast Biscuit
- Food Product F: White Bread (Experimental): White Bread
  Interventions: Other: Food Product F: White Bread

INTERVENTIONS:
Other: Reference Glucose
  Other Names: Glucose Standard (50g of Glucose)
  Arms: Reference Glucose
Other: Food Product A: Corn Flakes
  Other Names: Corn Flakes
  Arms: Food Product A: Corn Flakes
Other: Food Product B: Ginger Bread
  Other Names: Ginger Bread
  Arms: Food Product B: Ginger Bread
Other: Food Product C:Sandwiched Breakfast Biscuit
  Other Names: Sandwiched Breakfast Biscuit
  Arms: Food Product C:Sandwiched Breakfast Biscuit
Other: Food Product D: Crackers Nature
  Other Names: Crackers Nature
  Arms: Food Product D: Crackers Nature
Other: Food Product E: Breakfast Biscuit
  Other Names: Breakfast Biscuit
  Arms: Food Product E: Breakfast Biscuit
Other: Food Product F: White Bread
  Other Names: White Bread
  Arms: Food Product F: White Bread

SUMMARY:
The purpose of this study is to determine and compare the glycaemic index values and response parameters of 6 food products between 3 laboratories.

DETAILED DESCRIPTION:
This study will be performed at 3 centers and 15 subjects will be recruited at each center.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-35 years inclusive.
2. Non-smoker.
3. BMI 19.0-25.0 kg/m2 inclusive.
4. Healthy subjects with:

   * Fasting plasma glucose < 5,6 mM (ADA criteria,2011)
   * Insulin resistance index based on homeostasis model assessment (HOMA-IR) <1.70
   * Fasting lipids: triglyceride <1.70mmol/L, LDL-cholesterol<5.00 mmol/L and HDL-cholesterol >1.03mmol/L for males or >1.29mmol/L for females (IDF criteria for metabolic syndrome, 2006)
   * Gamma-GT, AST and ALT <1.5 times the upper limit of normal (ULN)
   * Complete blood count: Normal full blood count according to the investigator
   * Systolic blood pressure <130 mmHg
   * Diastolic blood pressure <85 mmHg
   * Resting heart rate 50-90 beats per minutes (after 3 minutes rest).
5. Stable dietary habits; normal eating patterns; no history of eating disorders or strict dieting.
6. Moderate level of physical activity (from basic daily activity to a high level of physical activity (regular physical activity at least 3 times per week))
7. Able to fast for at least 10 hours the night before each test session.
8. Able to refrain from eating legumes and drinking alcohol the day before each test session.
9. Subject covered by social security or covered by a similar system
10. Subject not taking any treatment for anorexia, weight loss, or any form of treatment likely to interfere with metabolism or dietary habits
11. Subject having given written consent to take part in the study

Exclusion Criteria:

1. Following a restrictive or specific diet.
2. Suffering from any inflammatory or metabolic diseases
3. Suffering from mental illness.
4. Suffering from any food allergies or hypersensitivities (wheat, milk, egg, nuts, etc).
5. Taking any regular prescription medication at the time of inclusion that should interfere with carbohydrate metabolism (except regular oral contraception medication, thyroid replacement therapy)
6. Female who is pregnant (positive test results), lactating, planning pregnancy or not using acceptable contraceptive.
7. Subject having taken part in another clinical trial within the last week.
8. Subject currently taking part in another clinical trial or being in the exclusion period of another clinical trial.
9. Subject undergoing general anaesthesia in the month prior to inclusion.
10. Subject in a situation which in the investigator's opinion could interfere with optimal participation in the present study or could constitute a special risk for the subject.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2013-06; Primary Completion 2013-11 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Determine and Perform Inter-Laboratory Comparison of Glycaemic Index Values of 6 Food Products | 0-120 minutes

SECONDARY OUTCOMES:
Determine and Perform Inter-Laboratory Comparison of Incremental Area Under the Curve (iAUC) of Glycaemia for Each of the 6 Food Products | 0-120 minutes
Determine and Perform Inter-Laboratory Comparison of the Glucose Cmax for Each of the 6 Food Products | 0-120 minutes
Determine and Perform Inter-Laboratory Comparison of the Blood Glucose Delta Peak for Each of the 6 Food Products | 0-120 minutes
Determine and Perform Inter-Laboratory Comparison of Insulinemic Index for Each of the 6 Food Products | 0-120 minutes
Determine and Perform Inter-Laboratory Comparison of the Incremental Area Under the Curve (iAUC) of Insulinemia for Each of the 6 Food Products | 01-20 minutes
Determination and Perform Inter-Laboratory Comparison of Insulin Cmax for Each of the 6 Food Products | 0-120 minutes
Determine and Perform Inter-Laboratory Comparison of the Blood Insulin Delta Peak for Each of the 6 Food Products | 0-120 minutes
Determine the Intra-Laboratory Variability for the iAUC of Glycaemia | 0-120 minutes
Determine the Intra-Laboratory Variability of the iAUC of Insulinemia | 0-120 minutes

CONTACTS AND LOCATIONS:
Overall Officials: David Gendre, Dr., Principal Investigator — BioFortis; Thomas Wolever, Dr., Principal Investigator — Glycemic Index Laboratories, Inc; Jennie Brand Miller, Dr., Principal Investigator — University of Sydney
Locations (3):
- Human Nutrition Unit, The University of Sydney, Sydney, Australia
- Glycemic Index Laboratories, Toronto, Ontario, Canada
- Biofortis, Saint-Herblain, France